CLINICAL TRIAL: NCT06104423
Title: Open-label, Multicenter, multinAtionaL, inteRventional Clinical Trial to Assess Efficacy and Safety of the exteMporaneous combInation of Nebivolol and Ramipril in hypertenSIve pAtients - ARTEMISIA Study
Brief Title: Open-label inteRventional Clinical Trial to Assess Efficacy and Safety of the exteMporaneous combInation of Nebivolol and Ramipril in hypertenSIve pAtients
Acronym: ARTEMISIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEIN/22/NeRam-Hyp/001; 2022-003060-25 (EudraCT Number)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Hypertension; Combination Therapy; Nebivolol; Ramipril; Fixed Dose Combination
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebivolol 5 mg (Active Comparator): MONOTHERAPY PERIOD 1 (4 weeks): Eligible patients entered a 4 weeks run-in period (week -4 to week 0) on the same day of the screening visit.
  Patients previously receiving Neb 5 mg continued the same treatment, while patients receiving any other BBs were switched to Neb 5 mg.
  COMBINATION THERAPY PERIOD 2 (12 weeks): During the Assessment period of 12 weeks (week 0_Baseline to week 12) uncontrolled patients will be treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients will continue with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg will be up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg. Controlled patients will continue same therapy.
  Interventions: Drug: Nebivolol 5 mg; Drug: Ramipril 2.5/5/10 mg
- Ramipril 2.5/5/10 mg (Active Comparator): MONOTHERAPY PERIOD 1 (4 weeks): Eligible patients entered a 4 week run-in (week -4 to week 0) period on the same day of the screening visit.
  Patients previously receiving RAM 5 mg continued the same treatment, while patients receiving any other ACE-i were switched to RAM 5 mg.
  COMBINATION THERAPY PERIOD 2 (12 weeks): During the Assessment period of 12 weeks (week 0_Baseline to week 12) uncontrolled patients will be treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients will continue with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg will be up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg. Controlled patients will continue same therapy.
  Interventions: Drug: Nebivolol 5 mg; Drug: Ramipril 2.5/5/10 mg

INTERVENTIONS:
Drug: Nebivolol 5 mg — 1 tablet of study medication (5mg) to be administered orally according to instructions of Investigator.
Drug: Ramipril 2.5/5/10 mg — 1 tablet of study medication (2.5mg or 5mg or 10mg) to be administered orally according to instructions of Investigator.

SUMMARY:
Open-label, inteRventional clinical Trial to assess EffIcacy and safety of the exteMporaneous combInation of Nebivolol and Ramipril in hypertenSIve pAtients.

DETAILED DESCRIPTION:
This is a Phase IV, interventional, multicenter, open-label, multinational study with 2 study periods (a Run-in period of 4 weeks and an Assessment period of 12 weeks) to assess the efficacy and safety of the extemporaneous combination of Nebivolol (NEB) and Ramipril (RAM) in reducing Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) in hypertensive patients uncontrolled by monotherapy.

The trial was conducted in 16 investigational clinical sites in Bulgaria, Poland, and Hungary.

Note: For the purpose of this study, uncontrolled blood pressure (BP) is defined as sitting SBP/DBP:

* ≥ 130/80 mmHg in patients < 65 years old
* ≥ 140/80 mmHg in patients ≥ 65 years old

Screening Visit 1 (Week -4):

Hypertensive patients with SBP ranging from ≥ 140 to ≤ 179 mmHg and/or DBP ranging from ≥ 90 to ≤ 109 mmHg on treatment, for at least 30 days prior to screening, with NEB 5 mg or any other Beta Blockers (BBs), or RAM 5 mg or any other Angiotensin-converting enzyme inhibitors (ACE-i) will be screened for eligibility (Visit1). Patients that did not meet eligibility criteria will be considered as screening failures and will not be re-screened.

Run-in period from Visit 1 (Week -4) to Visit 2 (Week 0):

On the same day of the Screening Visit, eligible patients will enter a Run-in period, during which:

* Patients receiving NEB 5 mg or RAM 5 mg will continue the same therapy for 4 weeks.
* Patients on any other BB will be assigned to monotherapy with NEB 5 mg while patients on any other ACE-i will be assigned to monotherapy with RAM 5 mg for 4 weeks. The study is designed in order to ensure that 1:1 ratio between patients in the NEB and RAM arms will be achieved.

Assessment period from Visit 2 (Week 0) to Visit 5 (Week 12):

After 4 weeks (± 2 days) of the Run-in period of monotherapy (Week 0), BP will be further assessed at Visit 2. Patients with uncontrolled BP levels (sitting BP ≥ 130/80 mmHg in patients < 65 years old/sitting BP ≥ 140/80 mmHg in patients ≥ 65 years old) at Visit 2, with adequate treatment adherence (ranging between 80% to 120%) and who did tolerate the treatment, will enter into the Assessment period and will be assigned to the extemporaneous combination of NEB/RAM 5/2.5 mg. Patients with controlled BP levels (sitting BP < 130/80 mmHg in patients < 65 years old/sitting BP < 140/80 mmHg in patients ≥ 65 years old) and/or who do not tolerate the treatment or have an adherence range below 80% or above 120%, will be withdrawn from the study (drop-out patients).

After 4 weeks ± 2 days in the Assessment period (Week 4), patients BP will be further evaluated at Visit 3: patients with controlled BP levels (sitting BP < 130/80 mmHg in patients < 65 years old/sitting BP < 140/80 mmHg in patients ≥ 65 years old) will continue the same extemporaneous combination, while patients with uncontrolled BP levels (sitting BP ≥ 130/80 mmHg in patients < 65 years old/sitting BP ≥ 140/80 mmHg in patients ≥ 65 years old) will be up-titrated from NEB/RAM 5/2.5 mg to NEB/RAM 5/5 mg for further 4 weeks ± 2 days.

After further 4 weeks ± 2 days (Week 8) the BP will be assessed again (Visit 4): controlled patients will continue the same extemporaneous combination, while uncontrolled patients:

* if on NEB/RAM 5/2.5 mg, will be up-titrated to NEB/RAM 5/5 mg for further 4 weeks

  ± 2 days (Visit 5, Week 12);
* if on NEB/RAM 5/5 mg, will be up-titrated to NEB/RAM 5/10 mg for further 4 weeks ± 2 days (Visit 5, Week 12).

At the end of the Assessment period (12 weeks ± 2 days), at Visit 5, the antihypertensive effect of the extemporaneous combination (NEB/RAM 5/2.5 mg, NEB/RAM 5/5 mg or NEB/RAM 5/10 mg) will be evaluated.

To correctly evaluate the additional effect of the combination therapy, the number of patients with uncontrolled BP on NEB or RAM monotherapy needs to be balanced at Visit 2. To maintain a 1:1 ratio during the Assessment period a cap of 110 patients for each treatment arm (i.e., NEB and RAM) will be included at Visit 2 to maintain a balanced number of uncontrolled patients entering the Assessment period for each drug.

The evaluation will be done every 50 patients. If the entrance in the Assessment period for 1 of the 2 tested drugs will deviate more than 5%, a corrective measure will be initiated: according to the enrollment site statistics, 1 or more sites will be informed to enroll a greater number of patients being treated with the least represented drug in the Assessment period.

ELIGIBILITY:
Inclusion Criteria:

Patient will be considered eligible to be enrolled in the study only if he/she meets all the following inclusion criteria:

1. Willing to comply with all study activities and procedures for the duration of the study and provided signed, written informed consent prior to any study procedures at Screening Visit.
2. Male or female patients aged ≥ 18 years with hypertension with mean sitting SBP ≥ 140 mmHg and ≤ 179 mmHg and/or mean sitting DBP ≥ 90 mmHg and

   ≤ 109 mmHg at Visit 1 (screening), while on monotherapy treatment either with BBs (NEB 5 mg or any dose if other BB) or ACE-is (RAM 5 mg or any dose if other ACE-i) for at least 30 days before Visit 1 (screening) and, as per Investigator's judgement, is deemed appropriate for a combination treatment with BB and ACE-i.
3. Ability to take oral medication and willing to adhere to the drug regimen.
4. Female patient of childbearing potential is eligible to participate if she is not pregnant, or not breastfeeding. A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile. Women of childbearing potential must agree to use of highly effective contraception (e.g., method of birth control throughout the study period and for 4 weeks after study completion defined as a method which results in a failure rate of less than 1% per year) and also must refrain from donating or storing eggs during this time. Highly effective contraception methods can be:

   * Combined hormonal contraception (estrogen- and progestogen-containing) associated with inhibition of ovulation (oral, intravaginal, and transdermal).
   * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, and implantable).
   * Intrauterine device.
   * Intrauterine hormone-releasing system.
   * Bilateral tubal occlusion.
   * Vasectomized partner (procedure conducted at least 2 months before the screening), (provided that partner is the sole sexual partner of the trial participant and that the vasectomized partner has received medical assessment of the surgical success).
5. A male patient must agree to use contraception during the whole study period and for at least 1 week after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

Any patient who meets any of the following criteria will not qualify for entry into the study:

1. Patients with documented history of hypersensitivity to NEB, RAM, other BBs or other ACE-is, or any related products, excipients of the formulations, as outlined in the relevant Investigator's Brochure (IB), summary of product characteristics (SmPC) or local package inserts for Nebivolol and Ramipril.
2. Patients with serious disorders (in the opinion of the Investigator) which may limit the ability to evaluate the efficacy or safety of the tested medications, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine, or metabolic, hematological, or oncological, neurological, and psychiatric diseases. The same applies for immunocompromised and/or neutropenic patients.
3. Patients having a history of the following conditions within the last 6 months:

   myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, bypass surgery, heart failure, hypertensive encephalopathy, valve replacement (transcatheter aortic valve implantation, mitraclip), cerebrovascular accident (stroke), or transient ischemic attack.
4. Patients with condition of hypotension with SBP < 90 mmHg and/or DBP < 60 mmHg.
5. Acute heart failure (12 months before enrolment), cardiogenic shock, or episodes of heart failure decompensation requiring intravenous inotropic therapy.
6. Patients with secondary hypertension of any etiology including renal diseases, Cushing's syndrome, hyperaldosteronism, renovascular disease and thyroid disorders.
7. Patients with severe heart failure (New York Heart Association classification III-IV) a narrowing of the aortic or bicuspid valve, an obstruction of cardiac outflow (obstructive, hypertrophic cardiomyopathy), obstruction of the outflow tract of the left ventricle (e.g., high grade aortic stenosis) or symptomatic coronary disease.
8. Patients with clinical evidence of renal disease (including significant bilateral renal artery stenosis or renal artery stenosis in a single functioning kidney), severe renal impairment or renal transplant.
9. Patients with clinically relevant hepatic impairment.
10. Patients with a history of angioneurotic edema.
11. Patients with sick sinus syndrome, including sino-atrial block.
12. Patient with second- and third-degree heart block (without a pacemaker).
13. History of bronchospasm and bronchial asthma.
14. Untreated phaeochromocytoma.
15. Patients with bradycardia (heart rate < 60 bpm; < 50 bpm in patients already on BBs treatment).
16. Patient with history of metabolic acidosis.
17. Patients with severe peripheral circulatory disturbances.
18. Participation in another interventional study within the last 30 days before Screening Visit (Visit 1).
19. Patients with diseases that, in the opinion of the Investigator, prevent a careful adherence to the protocol.
20. Patients using and not suitable for withdrawing the prohibited medications prior to the administration of study treatment.
21. Pregnant and breastfeeding women. NOTE: a pregnancy test will be performed on all women of childbearing potential at each study visit.
22. Patients with medical history of cirrhosis (Child Pugh class B or higher).
23. History of unexplained syncope within the prior 2 years, or a known syncopal disorder.
24. Patients who received renal denervation in the last 3 years or other device-based nonpharmacological treatment of hypertension.
25. Any other contraindication to either NEB or RAM as per respective SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovambattista Desideri, Prof, Principal Investigator — University of Roma La Sapienza
Locations (1):
- A & P Kft., Hosszúhetény, Hungary

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After Screening visit, eligible patients entered a 4 week run-in period (Monotherapy period from V1 week -4 to V2 week 0) on the same day of the screening visit. Patients receiving NEB 5 mg or RAM 5 mg will continue to receive the same, while patients on any other BBs or ACE-is, will receive NEB 5 mg or RAM 5 mg respectively prior to enrolment into the study.
  Assessment period (Combination therapy) starts from V2 week 0 (baseline) till V5 week 12 for a total of 12 weeks
Groups:
- Nebivolol 5 mg: MONOTHERAPY PERIOD 1 (4 weeks): Eligible patients entered a 4 weeks run-in period (week -4 to week 0) on the same day of the screening visit.
  Patients previously receiving Neb 5 mg continued the same treatment, while patients receiving any other BBs were switched to Neb 5 mg.
  Nebivolol 5 mg: 1 tablet of study medication (5mg) to be administered orally according to instructions of Investigator.
- Ramipril 5 mg: MONOTHERAPY PERIOD 1 (4 weeks): Eligible patients entered a 4 week run-in (week -4 to week 0) period on the same day of the screening visit.
  Patients previously receiving RAM 5 mg continued the same treatment, while patients receiving any other ACE-i were switched to RAM 5 mg.
  Ramipril 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
- Neb 5mg/ Ram 2.5, 5, 10 mg: COMBINATION THERAPY PERIOD 2 (12 weeks): During the Assessment period of 12 weeks (week 0 to week 12) uncontrolled patients will be treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients will continue with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg will be up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg. Controlled patients will continue same therapy. Nebivolol 5 mg: 1 tablet of study medication (5mg) to be administered orally according to instructions of Investigator. Ramipril 2.5/5/10 mg: 1 tablet of study medication (2.5mg or 5mg or 10mg) to be administered orally according to instructions of Investigator.
Period: MONOTHERAPY Period 1 RunIn (-4W to W0)
Arm/Group | Nebivolol 5 mg | Ramipril 5 mg | Neb 5mg/ Ram 2.5, 5, 10 mg
Started | 128 (Patients previously receiving NEB 5 mg continued the same treatment, while patients receiving any other Beta blocker were switched to NEB 5 mg.) | 138 (Patients previously receiving RAM 5 mg continued the same treatment, while patients receiving any other ACEi were switched to RAM 5 mg.) | 0
Completed | 124 | 131 | 0
Not Completed | 4 | 7 | 0
Not completed — Not compliant with eligibility criteria | 3 | 6 | 0
Not completed — Lab abnormal results | 1 | 1 | 0
Period: Combo Period 2 Assessment (W0 to W12)
Arm/Group | Nebivolol 5 mg | Ramipril 5 mg | Neb 5mg/ Ram 2.5, 5, 10 mg
Started (Number of subjects (Total 255) starting Combo Period 2 Assessment (W0 to W12) is not equal to the number completing the preceding monotherapy period (Total 266) because 11 patients were dropped before starting the combination phase. A total of 255 patients therefore started the combination phase with Neb/Ram 5/2.5 mg.) | 0 | 0 | 255 (All 255 patients in the combination phase were treated sequentially and started with Neb/Ram 5/2.5 mg.)
Completed the Study With Neb 5 mg/ Ram 2.5 mg | 0 | 0 | 85 (85 patients out of these 255 patients have maintained Neb 5/Ram 2.5 mg during all the assessment period 2 (Combination therapy period 2) from week 0 to week 12.)
Completed the Study With Neb 5 mg/ Ram 5 mg | 0 | 0 | 99 (All 255 patients in the combination phase were treated sequentially and started with Neb/Ram 5/2.5 mg. A total of 170 out of these 255 patients were uncontrolled at V3 and/or V4 and were therefore sequentially up-titrated to higher dosage(s): 99 patients were up-titrated to NEB/RAM 5/5 mg at Visit 3 (Week 4) or Visit 4 (Week 8) and have completed combination therapy with Neb 5/Ram 5mg.)
Completed the Study With Neb 5 mg/ Ram 10 mg | 0 | 0 | 71 (All 255 patients in the combination phase were treated sequentially and started with Neb/Ram 5/2.5 mg. A total of 170 out of these 255 patients were uncontrolled at V3 and/or V4 and were therefore sequentially up-titrated to higher dosage(s): 71 patients - after being firstly up-titrated to NEB/RAM 5/5 mg at Visit 3 (Week 4) - were subsequently up-titrated to NEB/RAM 5/10 mg at Visit 4 (Week 8) and have completed combination therapy with Neb 5/Ram 10mg.)
Completed | 0 | 0 | 255
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients(pts) were treated sequentially and only pts uncontrolled by lower dosage(s) were uptitrated to the higher ones. Specifically all pts N=255 in the Combo phase(W0 Baseline) started with NEB/RAM 5/2.5mg dose. Then, out of these 255pts, 85pts remained on NEB/RAM 5/2.5mg for the entire Combo period, whereas 99pts were uptitrated to NEB/RAM 5/5mg at V3(W4) or V4(W8) and 71pts - after being firstly uptitrated to NEB/RAM 5/5mg at V3(W4) - were subsequently uptitrated to NEB/RAM 5/10mg at V4(W8)
Groups:
- Nebivolol 5 mg/Ramipril 2.5 mg: COMBINATION THERAPY PERIOD (12 weeks): During the Assessment period of 12 weeks (week 0 to week 12) uncontrolled patients were treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg were up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients continued with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg were up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg were up-titrated to Ramipril 5 mg. Controlled patients continued same therapy.
  Nebivolol 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
  Ramipril 2.5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
- Nebivolol 5 mg/Ramipril 5 mg: COMBINATION THERAPY PERIOD (12 weeks): During the Assessment period of 12 weeks (week 0 to week 12) uncontrolled patients were treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg were up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients continued with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg were up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg were up-titrated to Ramipril 5 mg. Controlled patients continued same therapy.
  Nebivolol 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
  Ramipril 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
- Nebivolol 5 mg/Ramipril 10 mg: COMBINATION THERAPY PERIOD (12 weeks): During the Assessment period of 12 weeks (week 0 to week 12) uncontrolled patients were treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg were up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients continued with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg were up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg were up-titrated to Ramipril 5 mg. Controlled patients continued same therapy.
  Nebivolol 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
  Ramipril 10 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
- Total: Total of all reporting groups
Arm/Group | Nebivolol 5 mg/Ramipril 2.5 mg | Nebivolol 5 mg/Ramipril 5 mg | Nebivolol 5 mg/Ramipril 10 mg | Total
Number analyzed (Participants) | 85 | 99 | 71 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 63 | 72 | 60 | 195
  >=65 years | 22 | 27 | 11 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (12.45) | 55.7 (13.89) | 54.0 (11.59) | 55.1 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 41 | 37 | 133
  Male | 30 | 58 | 34 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 84 | 98 | 71 | 253
  Not Hispanic or Latino | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome: Change in Mean Sitting SBP
Description: To assess the antihypertensive efficacy of the extemporaneous combination of Nebivolol 5 mg in combination with Ramipril 2.5 mg or 5 mg or 10 mg in lowering the sitting systolic BP between Visit 2(Week 0) and Visit 5 (Week 12) in patients with uncontrolled BP previously treated with Nebivolol 5 mg or Ramipril 5 mg monotherapies for at least 4 weeks during run-in period.
Time Frame: 12 weeks of combination therapy treatment. From study Visit 2 (Week 0) to study Visit 5 (Week 12)
Population: All pts who signed ICF, met all criteria, received at least one dose of assigned treatment during RunIn, completed RunIn, met criteria at V2 (uncontrolled sitting BP≥130/80 mmHg in pts<65y old/ BP≥140/80 mmHg in pts≥65 y old atV2, with adequate treatment adherence 80-120%), tolerated treatment, had at least one dose of combination therapy and had at least baseline V2 and V5 assessments with primary efficacy data. 239 pts were included in Modified intention to treat for primary efficacy analysis
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Nebivolol 5 mg/Ramipril 2.5/5/10 mg: COMBINATION THERAPY PERIOD (12 weeks): During the Assessment period of 12 weeks (week 0 to week 12) uncontrolled patients will be treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients will continue with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg will be up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg. Controlled patients will continue same therapy.
  Nebivolol 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
  Ramipril 2.5/5/10 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
Arm/Group | Nebivolol 5 mg/Ramipril 2.5/5/10 mg
Number analyzed (Participants) | 239
mmHg | -19.2 (8.62)
Statistical Analysis 1: Comparison: Nebivolol 5 mg/Ramipril 2.5/5/10 mg; Primary endpoint, verified on the single cohort of patients who completed the monotherapy run-in period, is calculated as the mean difference in sitting systolic blood pressure between Visit 2 (Week 0, Baseline Visit of the combination therapy) and Visit 5 (Week 12, End of Study Visit). This is not a comparison of two different arms, but a comparison of two measurements taken from the same patient treated with combination therapy (single arm paired pre- vs. post-combination therapy comparison); Test type: Superiority; p < 0.001, paired t-test; Mean difference pre vs post treatment = -19.2, 95% CI 2-sided [-26.0 to -14.0], Standard Deviation 8.62

ADVERSE EVENTS:
Time Frame: From Informed Consent signature at screening visit (Visit 1) occurring 4 week previous than Baseline assessment (Week 0 - Visit 2) to last visit at Week 12 (Visit 5) for an average of 16 weeks. Furthermore patients having any ongoing Adverse Event/Serious Adverse Event at the end of the treatment (Week 12 - Visit 5), will be followed for further 2 weeks via a phone call to check about the status of the Adverse Events/Serious Adverse Events, extending the time frame to a total of 18 weeks.
Description: Safety Population(SP):All patients(pt) enrolled that received at least one dose of the assigned treatment during RunIn. One pt wasn't dosed wasn't part of SP. If a pt reports the same AE more than once within that System Organ Class SOC/Preferred Term PT, then that pt will be counted only once for that SOC or PT. For the purpose of safety analyses concerning the combination therapy period, 255, 170, and 71 patients were exposed to at least 1 dose of the NEB/RAM 5/2.5 mg,5 mg,10 mg, respectively.
Groups:
- Nebivolol 5 mg: MONOTHERAPY PERIOD (4 weeks): Eligible patients entered a 4 weeks run-in period (week -4 to week 0) on the same day of the screening visit.
  Patients previously receiving Neb 5 mg continued the same treatment, while patients receiving any other BBs were switched to Neb 5 mg.
  Nebivolol 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
- Ramipril 5 mg: MONOTHERAPY PERIOD (4 weeks): Eligible patients entered a 4 week run-in (week -4 to week 0) period on the same day of the screening visit.
  Patients previously receiving RAM 5 mg continued the same treatment, while patients receiving any other ACE-i were switched to RAM 5 mg.
  Ramipril 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
- Nebivolol 5 mg/Ramipril 2.5 mg: COMBINATION THERAPY PERIOD (12 weeks): During the Assessment period of 12 weeks (week 0 to week 12) uncontrolled patients will be treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients will continue with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg will be up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg. Controlled patients will continue same therapy.
  Nebivolol 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
  Ramipril 2.5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
- Nebivolol 5 mg/Ramipril 5 mg: COMBINATION THERAPY PERIOD (12 weeks): During the Assessment period of 12 weeks (week 0 to week 12) uncontrolled patients will be treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients will continue with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg will be up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg. Controlled patients will continue same therapy.
  Nebivolol 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
  Ramipril 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
- Nebivolol 5 mg/Ramipril 10 mg: COMBINATION THERAPY PERIOD (12 weeks): During the Assessment period of 12 weeks (week 0 to week 12) uncontrolled patients will be treated with the extemporaneous combination of Nebivolol 5 mg and Ramipril 2.5 mg for 4 weeks. Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg in uncontrolled patients for further 4 weeks while controlled patients will continue with Nebivolol 5 mg/Ramipril 2.5 mg therapy. After 8 weeks Ramipril 5 mg will be up-titrated to Ramipril 10 mg in the uncontrolled patients as well as Ramipril 2.5 mg will be up-titrated to Ramipril 5 mg. Controlled patients will continue same therapy.
  Nebivolol 5 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
  Ramipril 10 mg: 1 tablet of study medication to be administered orally according to instructions of Investigator.
Arm/Group | Nebivolol 5 mg | Ramipril 5 mg | Nebivolol 5 mg/Ramipril 2.5 mg | Nebivolol 5 mg/Ramipril 5 mg | Nebivolol 5 mg/Ramipril 10 mg
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/138 | 0/255 | 0/170 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/138 | 0/255 | 1/170 | 0/71
Other Adverse Events (participants affected / at risk) | 0/128 | 0/138 | 14/255 | 18/170 | 6/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebivolol 5 mg (N=128) | Ramipril 5 mg (N=138) | Nebivolol 5 mg/Ramipril 2.5 mg (N=255) | Nebivolol 5 mg/Ramipril 5 mg (N=170) | Nebivolol 5 mg/Ramipril 10 mg (N=71)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebivolol 5 mg (N=128) | Ramipril 5 mg (N=138) | Nebivolol 5 mg/Ramipril 2.5 mg (N=255) | Nebivolol 5 mg/Ramipril 5 mg (N=170) | Nebivolol 5 mg/Ramipril 10 mg (N=71)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid 19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT06104423/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT06104423/SAP_001.pdf